CLINICAL TRIAL: NCT00933127
Title: Association of FC-Gamma Receptor Genotypes With Response and Clinical Benefit With Addition of Rituximab to CHOP Chemotherapy in Patients With Follicular Lymphoma (FL)
Brief Title: S8809-S9800-S9911-S9704-A Study of Blood and Tissue Samples From Patients With Follicular Lymphoma Treated With Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride, Vincristine, and Prednisone
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000630578; SWOG-S8809-S9800-S9911-S9704-A
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood and tissue samples from patients with follicular lymphoma treated with rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test for association of polymorphisms in Fc-gamma (Fcγ) receptors IIa (H/R131) and IIIa (V/F158) with progression-free survival and clinical response in patients with follicular non-Hodgkin lymphoma treated with rituximab and CHOP chemotherapy comprising cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone.
* To assess novel polymorphisms in Fcγ receptors for predictive and prognostic significance in patients treated with this regimen.

OUTLINE: Genomic DNA extracted from paired samples of serum and formalin-fixed paraffin-embedded tissue is analyzed for R131H polymorphism in Fcγ receptor IIa and V158F polymorphism in Fcγ receptor IIIa by TaqMan-based assay. The DNA is also analyzed for genotypes corresponding with several other polymorphisms in Fcγ receptors, as determined by the HapMap project. The resulting Fcγ receptor genotypes are then compared with clinical data from the Southwest Oncology Group database to identify associations between particular genotypes and progression-free survival, overall response, and complete response. A multivariate analysis incorporating clinical prognostic variables (e.g., age, stage, serum LDH level, extranodal disease, and performance status) is also performed to determine whether Fcγ receptor polymorphisms are independent predictive or prognostic markers for clinical outcome.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of follicular lymphoma
* Meets either of the following criteria:

  * Previously enrolled on clinical trial SW0G-8809 and treated with chemotherapy alone

    * Excess tissue sections available
  * Previously enrolled on clinical trial SWOG-9800 or SWOG-9911 and treated with a combination of chemotherapy and monoclonal antibody therapy
* Matched serum and tissue samples available from the SWOG Lymphoma Bank

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled to S8809 S9800 S9911 S9704 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Association of Fc-gamma (Fcγ) receptor genotypes with overall and/or progression-free survival and clinical response | retrospectively
Novel polymorphisms in Fcγ receptors for predictive and prognostic significance | retrospectively

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rimsza, MD, Study Chair — University of Arizona

REFERENCES:
- [Result] Persky DO, Dornan D, Goldman BH, Braziel RM, Fisher RI, Leblanc M, Maloney DG, Press OW, Miller TP, Rimsza LM. Fc gamma receptor 3a genotype predicts overall survival in follicular lymphoma patients treated on SWOG trials with combined monoclonal antibody plus chemotherapy but not chemotherapy alone. Haematologica. 2012 Jun;97(6):937-42. doi: 10.3324/haematol.2011.050419. Epub 2012 Jan 22. PMID 22271896